CLINICAL TRIAL: NCT02551900
Title: A Comparison of the Effect of Warm and Cold Water Exercise Training on Vascular Function in Type 2 Diabetic Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chulalongkorn University (Other)
Responsible Party: Principal Investigator, Assoc. Prof. Dr.Daroonwan Suksom, Faculty of Sport Science, Chulalongkorn University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SPSC-4
Record Dates: First submitted 2015-09-15; First posted 2015-09-16 (Estimated); Last update posted 2018-04-04 (Actual); Status verified 2018-04

CONDITIONS: Type 2 Diabetes
Keywords: Type 2 Diabetes; Vascular Function; Water Exercise; Warm Water; Cold Water
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (2):
- Warm water exercise & Cold water exercise (Experimental)
  Interventions: Other: Warm water exercise; Other: Cold water exercise
- Warm water exercise & Land cycling exercise (Active Comparator)
  Interventions: Other: Warm water exercise; Other: Land based cycling exercise

INTERVENTIONS:
Other: Warm water exercise — Warm water based cycling exercise training program will be based on cycling in warm water (temperature 34◦C ). Warm water exercise will be conducted at moderate intensity (60-70% maximum heart rate). The three groups were exercise 15 minutes on the first month, second month will be increased to 20 minutes and the last month will be increased to 30 minutes. The training program will be performed 3 times per week for 12 weeks.
Other: Cold water exercise — Cold water based cycling exercise training will be based on cycling in cold water (temperature 20◦C ). Cold water exercise will be conducted at moderate intensity (60-70% maximum heart rate). The three groups were exercise 15 minutes on the first month, second month will be increased to 20 minutes and the last month will be increased to 30 minutes. The training program will be performed 3 times per week for 12 weeks.
  Arms: Warm water exercise & Cold water exercise
Other: Land based cycling exercise — Land based cycling exercise training will be based on ride a bicycle ergometer (Monark 894e, Sweden). Land based cycling exercise training will be conducted at moderate intensity (60-70% maximum heart rate). The three groups were exercise 15 minutes on the first month, second month will be increased to 20 minutes and the last month will be increased to 30 minutes. The training program will be performed 3 times per week for 12 weeks.
  Arms: Warm water exercise & Land cycling exercise

SUMMARY:
Warm water based cycling exercise training would more favorable than cold water based cycling exercise training and land based cycling exercise in vascular function in type 2 diabetic patients.

ELIGIBILITY:
Inclusion Criteria:

* The inclusion criteria included type 2 diabetes (as defined by the American Diabetes Association), a baseline glycosylated hemoglobin (HbA1c) value of 7-9%, and no previous exercise training in the past 6 months. All participants were free from diabetic nephropathy, diabetic retinopathy, severe diabetic neurophathy, severe cardiovascular and cerebrovascular diseases.

Exclusion Criteria:

* Participants were excluded if they dropped out or completed less than 80% of the training schedule.

Ages: 60 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2014-09-01; Primary Completion 2015-09-15 (Actual); Study Completion 2016-12-15 (Actual)

PRIMARY OUTCOMES:
Change from baseline in glycemic control | Baseline, 12 weeks
  The glycemic control will be quantified using blood samples. Fasting blood glucose, HbA1c, insulin, homeostasis model assessment of insulin resistance (HOMA-IR) and C-reactive protein will be measured with standard procedures at the clinical laboratory (N health Lab, Samitivej, Sriracha, Thailand). Homeostasis model assessment (HOMA-IR will be calculated by using equation of [Fasting glucose (mg/dL) × Insulin level (uU/mL) / 405].
Change from baseline in vascular reactivity | Baseline, 12 weeks
  Vascular reactivity or brachial and popliteal artery flow-mediated dilatation (FMD) will be assessed with the ultrasound equipment (CX50, Philips, USA), using the blood occlusion technique on the right forearm and lower leg. The brachial artery and the popliteal artery will be imaged above the antecubital fossa in the longitudinal plane and proximal slightly above the popliteal fossa. Brachial FMD will be measured at baseline and the cuff placed around the right forearm will be inflated to 50 mmHg above systolic blood pressure for 5 minutes and then deflated for 5 minutes of recovery. While popliteal FMD will be measured at baseline and the cuff will be positioned on the lower right leg below the knee will be inflated to 250 mmHg for 5 minutes and then deflated for 5 minutes of recovery. FMD will be calculated from the formula FMD= (D2-D1)x100/D1 when D1 is the brachial or popliteal artery diameter at baseline, D2 is the maximal post-occlusion brachial or popliteal artery diameter.
Change from baseline in cutaneous blood flow | Baseline, 12 weeks
  Cutaneous blood flow will be determined by laser Doppler Flowmetry (DRT4, Moore Instrument, UK). Laser Doppler Flowmetry probes will be attached to the dorsum of middle fingertip and the dorsum of the foot. The occlusion cuffs will be placed around left middle upper arm and calf were inflated to a pressure of 50 mmHg above the systolic pressure and will be remained inflated for 3 minutes, after which it will be rapidly released, producing a brief high-flow state resulting in artery dilation due to increase shear stress. The peak Laser Doppler Flux (peak LDF) and after 5 min occlusion period will be recorded.

SECONDARY OUTCOMES:
Change from baseline in physical fitness | Baseline, 12 weeks
  Body composition will be measured using Body Composition Analyzer (Tanita BC-533, Japan)
Change from baseline in physical fitness | Baseline, 12 weeks
  Lower muscle strength will be measured with leg dynamometer (Tokyo, Japan).
Change from baseline in physical fitness | Baseline, 12 weeks
  Maximal oxygen consumption (VO2peak) will be assessed by bicycle ergometer (Monark: 824e, Sweden). Initial work load was 50 watt and increased stepwise by 25 W every 2 minutes (as measured using respiratory gas analyzer: Metamax 3B, Germany) until the subjects were no longer able to continue exercising.
Change from baseline in physical fitness | Baseline, 12 weeks
  Pulmonary function will be measured by spirometer ((MIR-Spirobank G)
Change from baseline in blood chemistry | Baseline, 12 weeks
  Nitric oxide (NO) will be measured in plasma samples with the commercial assay kit (Colorimetric nitric oxide assay kit, PromoKine, Germany).
Change from baseline in blood chemistry | Baseline, 12 weeks
  Malondialdehyde (MDA) will be determined using thiobarbituric acid reaction.
Change from baseline in blood chemistry | Baseline, 12 weeks
  C-reactive protein will be measured with standard procedures at the clinical laboratory (N health Lab, Samitivej, Sriracha, Thailand).
Change from baseline in Peripheral arterial stiffness | Baseline, 12 weeks
  Pulse wave velocity (brachial-ankle PWV) measurement will be assessed using Omron Colin VP1000 for measuring.

CONTACTS AND LOCATIONS:
Overall Officials: Daroonwan Suksom, Ph.D., Principal Investigator — Faculty of Sport Science Chulalongkorn University
Locations (1):
- Laemchabang stadium, Sukhumvit Rd, Si Racha, Changwat Chon Buri, Thailand